CLINICAL TRIAL: NCT00002053
Title: A Double-Blind Placebo-Controlled Group Comparative Study To Evaluate the Safety and Effectiveness of Aerosol Pentamidine in the Prophylaxis of Pneumocystis Carinii Pneumonia in Patients With AIDS Post First Episode PCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisons (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 022B; 87-72
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Pentamidine; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Pentamidine

INTERVENTIONS:
Drug: Pentamidine isethionate

SUMMARY:
To evaluate and compare the safety, tolerability, and efficacy of biweekly administration of aerosol pentamidine versus placebo when used as a prophylactic agent in patients who have recovered from their first episode of AIDS-associated Pneumocystis carinii pneumonia (PCP).

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT). If AZT is started during the study, patients must have received = or > 15 days of aerosol pentamidine before beginning AZT.

Prior Medication:

Allowed:

* Zidovudine (AZT). If AZT began prior to study entry, patients must have received = or > 15 days of AZT before beginning aerosol pentamidine.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Requiring ongoing active therapy for an opportunistic infection (O.I.) at time of entry or those with either of the following AIDS-defining O.I.'s prior to entry:
* Toxoplasmosis.
* Cryptococcosis.
* Transfusion dependent (requiring blood transfusion more than once per month). The last transfusion cannot have been given within 7 days of study entry.
* Pulmonary Kaposi's sarcoma (KS).
* Uncontrolled asthma.
* Active therapy for tuberculosis.

Patients with the following are excluded:

* Requiring ongoing active therapy for an opportunistic infection (O.I.) at time of entry or those with either of the following AIDS-defining O.I.'s prior to entry:
* Toxoplasmosis.
* Cryptococcosis.
* Transfusion dependent (requiring blood transfusion more than once per month). The last transfusion cannot have been given within 7 days of study entry.
* Pulmonary Kaposi's sarcoma (KS).
* Uncontrolled asthma.

Prior Medication:

Excluded within 30 days of study entry:

* Antiretroviral agents other than zidovudine (AZT).
* Immunomodulating agents.
* Corticosteroids.

Active therapy for tuberculosis.

Patients must:

* Have AIDS and recovered from their first episode of Pneumocystis carinii pneumonia (PCP).
* Be at least 2 weeks and no more than 24 weeks status post therapy for acute PCP.
* Have positive antibody to HIV by a Government-approved ELISA test kit, or confirmed Western blot test.
* Adequate pulmonary function (vital capacity = or > 80 percent of predicted; forced expiratory volume (FEV), 1 s = or > 65 percent of total FEV; and corrected pulmonary diffusion capacity > 60 percent of predicted).
* Free of acute medical problems.

Active substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Fisons Corp, Rochester, New York, United States

REFERENCES:
- [Background] Montaner JS, et al. Aerosolized pentamidine for the secondary prophylaxis of Pneumocystis carinii pneumonia in the acquired immunodeficiency syndrome: a report from the Canadian cooperative trial. Int Conf AIDS. 1989 Jun 4-9;5:295 (abstract no TBP54)